CLINICAL TRIAL: NCT05630924
Title: Children's Lifestyle, Diet, and Exercise Intervention - CHILDREN's Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not meeting recruitment targets
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Sesame Workshop (Unknown)
Responsible Party: Principal Investigator, Valentin Fuster, President of Mount Sinai Heart and Chairman, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 20-0655
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Healthy Lifestyle; Cardiovascular Health
Keywords: Children; Lifestyle; School-based Intervention; Cardiovascular Health; Health Promotion; Habits
MeSH Terms: conditions — Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SI! Program-NYC Children (Experimental): Receives 4 month health promotion educational intervention.
  Interventions: Other: SI! Program-NYC
- NYC Elementary School Children (No Intervention): The control group will be participating school children not enrolled in the program

INTERVENTIONS:
Other: SI! Program-NYC — SI! Program-NYC incorporates a comprehensive and integrated vision of CV health promotion that encompasses four (4) basic and interrelated components: body and heart, physical activity healthy diet; and emotional management.
  Arms: SI! Program-NYC Children

SUMMARY:
Cluster randomized trial to evaluate the impact of a health promotion intervention (the SI! - Program NYC) on the adapted Ideal Cardiovascular Health score (aICH) in children enrolled in New York City elementary schools.

DETAILED DESCRIPTION:
Cluster randomized trial to evaluate the impact of a health promotion intervention (the SI! - Program NYC) on the adapted Ideal Cardiovascular Health score (aICH) in children enrolled in New York City elementary schools. This study will enroll children of ages 5 to 6 and teachers from participating schools. Participating schools will be randomized to an intervention group or a control (non-intervention group). The SI! Program intervention will incorporate a comprehensive vision of cardiovascular health promotion that encompasses four basic components: body and heart, physical activity, healthy diet, and emotional management. The intervention will take place at baseline and a reintervention will take place at 2 years-follow up. The research team will assess an adapted version of the Ideal Cardiovascular Health (aICH) score (that includes body-mass-index Z-score, physical activity, diet, sleep time and smoking exposure) and the Knowledge, Attitudes, and Habits (KAH) score. The aICH will be evaluated at baseline, 2 years and 4 years follow-up; the KAH will be evaluated at baseline and after the first intervention, and prior and after the second intervention. The research team will also study the influence of factors in parents (socioeconomic and health-related variables), teachers (stress, teaching motivation, and health status), and the environment (pollution, housing, and neighborhood conditions) through parent/caregiver questionnaires, teacher questionnaires, publicly available data, and pollution data sourced from NASA satellites.

ELIGIBILITY:
Inclusion Criteria:

* NYC Elementary school Kindergarten Children
* Parents and teachers of participating children

Exclusion Criteria:

* Children who are Wards of the State
* Children or parents who cannot provide legally effective consent

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1294 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Adapted Ideal Cardiovascular Health Score (ICH) | Baseline
  The adapted ideal cardiovascular health score (ICH) includes 5 components: body-mass-index Z-score, physical activity, diet, sleep/screen time, and passive smoking status. The score will be calculated for five factors on a 0 to 100 scale, according to pre-defined, age adjused cut-offs recommended by the American Heart Association. Higher values represent better health outcomes.
Adapted Ideal Cardiovascular Health Score (ICH) | 2 years
  The adapted ideal cardiovascular health score (ICH) includes 5 components: body-mass-index Z-score, physical activity, diet, sleep/screen time, and passive smoking status. The score will be calculated for five factors on a 0 to 100 scale, according to pre-defined, age adjused cut-offs recommended by the American Heart Association. Higher values represent better health outcomes.
Adapted Ideal Cardiovascular Health Score (ICH) | 4 years
  The adapted ideal cardiovascular health score (ICH) includes 5 components: body-mass-index Z-score, physical activity, diet, sleep/screen time, and passive smoking status. The score will be calculated for five factors on a 0 to 100 scale, according to pre-defined, age adjused cut-offs recommended by the American Heart Association. Higher values represent better health outcomes.

SECONDARY OUTCOMES:
Knowledge, Attitudes, and Habits Score | Baseline
  Questionnaires will be given to assess the knowledge (K), attitudes (A) and habits (H) of the children representing each of the components of the intervention (KAH-diet, KAH-physical activity, and KAH-human body). An overall score representing the intervention as a whole (overall KAH) will be derived from the 39 items, ranging from 0-80. The overall KAH score is derived from the sum of each component-specific score (Diet, 0 to 30 points; Physical activity, 0 to 30 points; and Human body, 0 to 20 points).
Knowledge, Attitudes, and Habits Score | 4 months
  Questionnaires will be given to assess the knowledge (K), attitudes (A) and habits (H) of the children representing each of the components of the intervention (KAH-diet, KAH-physical activity, and KAH-human body). An overall score representing the intervention as a whole (overall KAH) will be derived from the 39 items, ranging from 0-80. The overall KAH score is derived from the sum of each component-specific score (Diet, 0 to 30 points; Physical activity, 0 to 30 points; and Human body, 0 to 20 points). Higher scores indicate better health outcomes.
Knowledge, Attitudes, and Habits Score | 2 years
  Questionnaires will be given to assess the knowledge (K), attitudes (A) and habits (H) of the children representing each of the components of the intervention (KAH-diet, KAH-physical activity, and KAH-human body). An overall score representing the intervention as a whole (overall KAH) will be derived from the 39 items, ranging from 0-80. The overall KAH score is derived from the sum of each component-specific score (Diet, 0 to 30 points; Physical activity, 0 to 30 points; and Human body, 0 to 20 points). Higher scores indicate better health outcomes.
Knowledge, Attitudes, and Habits Score | 2 years and 4 months
  Questionnaires will be given to assess the knowledge (K), attitudes (A) and habits (H) of the children representing each of the components of the intervention (KAH-diet, KAH-physical activity, and KAH-human body). An overall score representing the intervention as a whole (overall KAH) will be derived from the 39 items, ranging from 0-80. The overall KAH score is derived from the sum of each component-specific score (Diet, 0 to 30 points; Physical activity, 0 to 30 points; and Human body, 0 to 20 points). Higher scores indicate better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available to external researchers upon request after approval with a signed data sharing agreement
Supporting Information: SAP, ICF, CSR
Time Frame: Starting 9 months after publication
Access Criteria: Research team will respond with any requests to share IPD.